CLINICAL TRIAL: NCT05776303
Title: Phase II (Intervention): Good Bowls: Empowering Communities to Achieve Good Food Access and Health Equity
Brief Title: Good Bowls: Eat Well At Work
Acronym: EWAW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Equiti Food, LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); University of North Carolina, Chapel Hill (Other); University of North Carolina, Greensboro (Other); North Carolina State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-2412
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Nutrition, Healthy; Behavior, Eating
Keywords: Med-South Diet; Worksite Intervention; Subsidized Food; App-based Messaging
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Randomize 240 individuals in 8-10 worksites to either Good Bowls alone or Good Bowls + Phone App nudges at a 1:1 allocation ratio. Initial assignment will be followed for four months, after which the groups will crossover for the subsequent four months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Good Bowls + App Nudges, followed by Good Bowls alone (Experimental): Participants in this arm will be exposed to Good Bowls + App Nudges throughout the first four months followed by four months of Good Bowls alone.
  Interventions: Behavioral: Good Bowls; Behavioral: Good Bowls + App Nudges
- Good Bowls, followed by Good Bowls + App Nudges (Active Comparator): Participants in this arm will be exposed to Good Bowls alone throughout the first four months followed by four months of Good Bowls + App Nudges.
  Interventions: Behavioral: Good Bowls; Behavioral: Good Bowls + App Nudges

INTERVENTIONS:
Behavioral: Good Bowls — Healthy, frozen subsidized meals are made conveniently available on worksites.
Behavioral: Good Bowls + App Nudges — Healthy, frozen subsidized meals are made conveniently available on worksites.
  Additionally, Bluetooth enabled beacons will be set up at each worksite that will send location specific messages to an individual's Smartphone via an App. These messages will include nutritional information, tips, and behavioral nudges.

SUMMARY:
The goal of this clinical trial is to improve the health of workers at their worksite by providing subsidized healthy meals supported by nutrition education and behavioral nudges using mobile health and Bluetooth technology.

The aim of this study is to:

Randomize 240 individuals in 8-10 worksites to either Good Bowls alone or Good Bowls + Phone App nudges. Using a crossover design, the primary outcome is the score on a validated Mediterranean diet screener, with secondary outcomes including weight, blood pressure, carotenoid levels, and food security.

Participants: Workers at blue and white-collar worksites.

Procedures: Workers will be recruited from 8-10 worksites who will be initially randomized within each site to Good Bowls alone or Good Bowls + Phone App nudges. Initial assignment will be followed for four months, after which the groups will crossover for the subsequent four months. The investigators will collect survey data as well as some physiologic measures including skin scanning (non-invasive), weight, and blood pressure. Effects between groups will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Employed at participating worksite
* No plans to move from the area for at least 1 year
* Free living to the extent that participant has control over dietary intake
* Willing and able to provide written informed consent and participate in all study activities

Exclusion Criteria:

* Severe food allergies
* Advanced kidney disease (estimated creatinine clearance < 30 ml/min)
* Known psychosis or major psychiatric illness that prevents participation with study activities
* Cognitive impairment, frailty, or other disability such that individual cannot fully participate in study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in nutrition as measured by the Mediterranean Diet 14-Item Screener Score | Baseline, 4 months
  A slightly adapted version of the Mediterranean Diet 14-item validated screener will be used for nutritional assessment. The score ranges from 0-14, with a higher score indicating higher adherence to the Mediterranean Diet.
Change in nutrition as measured by the Mediterranean Diet 14-Item Screener Score | 4 months, 8 months
  A slightly adapted version of the Mediterranean Diet 14-item validated screener will be used for nutritional assessment. The score ranges from 0-14, with a higher score indicating higher adherence to the Mediterranean Diet.
Change in nutrition as measured by the Mediterranean Diet 14-Item Screener Score | Baseline, 8 months
  A slightly adapted version of the Mediterranean Diet 14-item validated screener will be used for nutritional assessment. The score ranges from 0-14, with a higher score indicating higher adherence to the Mediterranean Diet.

SECONDARY OUTCOMES:
Change in weight | Up to 8 months
  Weight in pounds as measured by electronic scale as the average of two measures. SECA 874dr scales will be used and assessed with standardized weights monthly for accuracy.
  Assessed at baseline (i.e., pre-intervention), 4 months (i.e., before crossover), 8 months (i.e., post-intervention).
Change in blood pressure | Up to 8 months
  Blood pressure (systolic and diastolic in mmHg) as measured by non-invasive automated monitor (Omron HEM-907XL, Vernon Hills, IL) with a first measure after seated for 5 minutes and 2 repeat measures at 1-minute intervals.
  Assessed at baseline (i.e., pre-intervention), 4 months (i.e., before crossover), 8 months (i.e., post-intervention).
Change in skin carotenoids | Up to 8 months
  Skin carotenoids as measured by a Reflection Spectroscopy Device ("Veggie Meter"™) placed on the participant's finger for a simple scan for three separate trials. Scores range from 0-800 arbitrary units with higher estimated value indicating greater carotenoid concentrations.
  Assessed at baseline (i.e., pre-intervention), 4 months (i.e., before crossover), 8 months (i.e., post-intervention).
Change in food security | Up to 8 months
  Food security as measured by the 2-Item Food Security Screening Tool. The two item response categories are: "Often True," "Sometimes True," "Never True" or "Don't Know" for the past 12 months. Often true and sometimes true are categorized as food insecure.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Ribisl, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University ofNorth Carolina (UNC) and Equiti Foods, LLC.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator with IRB, IEC, or REB approval and an executed data use agreement with UNC and Equiti Foods, LLC